CLINICAL TRIAL: NCT07284329
Title: Examining the Efficacy of a Parent-targeted Co-designed Digital Media Intervention to Increase Recruitment Rates Across a Multi-site Randomized Clinical Trial in Canadian NICU's
Brief Title: Examining the Efficacy of a Digital Media Intervention to Increase Recruitment Rates
Acronym: WHEAT-Boost
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Balpreet Singh, Associate Professor, Neonatologist, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1027137 (SWAT); CTR-184893/ CT1-184892 (Other Grant/Funding Number: ACT/CIHR)
Record Dates: First submitted 2025-11-19; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Consent Process
Keywords: Consent; Neonatal research; Family questionnaires; Digital media; Co-design; Study video
MeSH Terms: interventions — Methods; Videotape Recording

STUDY DESIGN:
Intervention Model Description: This study uses a stepped-wedge cluster randomized design, where participating NICU sites transition sequentially from the control (usual consent process) to the intervention (usual process plus digital media video) at randomized time points. Individual participants are exposed to only one condition based on the timing of their enrollment, making the study function as a parallel assignment design at the participant level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No-Video) Arm (No Intervention): Participants receive the standard informed consent or opt-out consent documentation for the WHEAT International Trial without any additional digital media support. Research staff approach parents/primary caregivers using the usual verbal and paper-based consent process. Families then complete a brief questionnaire about their understanding and experience with the consent process.
- Intervention (Video) Arm (Experimental): Participants receive the usual informed consent or opt-out consent documentation plus access to a co-designed 3.5-4-minute digital media video that explains the importance of neonatal research and key trial details in an accessible format. The video is intended to supplement and clarify the consent process to improve understanding and recruitment.
  Research staff provide parents/primary caregivers with a QR code linking to the video hosted on the WHEAT International Trial website. Families are encouraged to watch the video on their personal devices or hospital devices if needed. This is provided alongside the usual consent documentation during the NICU stay. Following this, families complete the same brief questionnaire about their experience and comprehension.
  Interventions: Behavioral: Intervention (Video) Arm

INTERVENTIONS:
Behavioral: Intervention (Video) Arm — A 3.5-4-minute co-designed digital media video created to supplement the standard consent process for the WHEAT International Trial.
  Arms: Intervention (Video) Arm

SUMMARY:
WHEAT-Boost is a Study Within A Trial (SWAT) that aims to improve how families are recruited into neonatal research studies by testing a new way of sharing information. The study is embedded within the larger WHEAT International Trial, a randomized clinical trial being conducted in Neonatal Intensive Care Units (NICUs) across Canada. The WHEAT International Trial investigates the best way to manage feeding around the time of blood transfusions in very premature infants (born before 30 weeks of pregnancy).

Recruiting families for research in the NICU is challenging. Parents are often stressed, overwhelmed, and unfamiliar with how clinical trials work, which can make it hard for them to process complex medical information and decide whether to take part. Traditional consent methods, such as paper forms, may not be enough to ensure families feel informed and comfortable with participation.

To address this, WHEAT-Boost will test whether adding a short, co-designed digital video helps improve recruitment rates. The video is 3.5 to 4 minutes long, available in English and French (with subtitles in other commonly spoken languages), and explains the importance of NICU research and details of the WHEAT International Trial in a simple and visual way. The video was co-developed with parents who have experience in the NICU to ensure the information is relevant and easy to understand.

NICU sites participating in the WHEAT Trial will be randomly assigned, in a stepped-wedge design schedule, to either continue using their usual recruitment methods, or to add the digital video to their recruitment approach. Parents in both groups will be asked to complete a short, voluntary questionnaire about their experience with the consent process and their understanding of the trial.

The main goal of WHEAT-Boost is to see if the video increases the number of families who agree to take part in the WHEAT Trial (known as the "opt-in rate"). The study will also look at whether the video reduces the number of families who later withdraw from the trial, and whether it improves parents' understanding of the study and their satisfaction with how information was shared.

If successful, the video could be used in other NICUs or future studies to help make research more accessible and inclusive for families. This approach could lead to stronger participation in neonatal trials, better-informed decisions by parents, and faster progress in improving care for premature babies.

DETAILED DESCRIPTION:
WHEAT-Boost is a stepped-wedge cluster randomized SWAT embedded within the ongoing WHEAT International Trial (NCT05213806), which evaluates feeding practices around blood transfusion in preterm infants. The SWAT aims to examine whether the addition of a co-designed digital media intervention improves recruitment outcomes, parental comprehension, and satisfaction with the research consent process in the NICU setting.

Fifteen Canadian NICUs participating in the WHEAT International Trial will be randomized in a stepped-wedge design to transition from the control condition (usual recruitment approach) to the intervention condition (usual approach plus video). Each site will act as its own control, with transitions occurring at 29-day intervals. All sites will begin in the control arm, using standard informed or opt-out consent materials, and then sequentially implement the video intervention according to the randomized schedule.

The intervention consists of a 3.5- to 4-minute digital video co-developed with a parent-partner advisory group. The video uses accessible language, storytelling, and visual elements to highlight the role and value of neonatal research and to clarify key details of the WHEAT Trial. It is delivered via a QR code linked to a secure website, enabling families to view the content on personal or institutional devices. The co-design approach ensures the material is tailored to the needs and concerns of NICU families, many of whom may experience emotional distress and information overload during their infant's hospitalization.

This SWAT will evaluate several outcomes. The primary outcome is the WHEAT Trial opt-in rate, defined as the proportion of eligible families who consent to enroll their infant in the trial. Secondary outcomes include the post-randomization withdrawal rate, parental comprehension of trial-specific information, and overall experience with the consent process. These will be measured using a brief questionnaire co-designed with the parent group and administered to all approached families, regardless of group assignment.

Analysis of the primary and secondary outcomes will follow intention-to-treat principles and will use generalized linear mixed models appropriate for the stepped-wedge design. Models will include random intercepts for sites and fixed effects for time and intervention status. For qualitative data from open-ended survey responses, an inductive thematic analysis approach will be applied.

This SWAT addresses a critical need for evidence-based strategies to enhance trial recruitment in high-stress clinical environments like the NICU. By supplementing conventional consent procedures with engaging, accessible media, the study seeks to normalize research participation and support informed decision-making by parents of vulnerable infants. If effective, this low-cost, scalable intervention could be readily adapted to other trials and clinical settings, advancing broader efforts to improve inclusivity and transparency in neonatal research.

ELIGIBILITY:
Inclusion Criteria (applied to infants/participants in WHEAT Trial):

Infant meets eligibility criteria for the WHEAT International Trial

Infant is <30 weeks gestational age at birth

Infant is admitted to one of the participating Canadian NICU sites

Parent(s)/primary caregiver(s) are approached for consent to participate in the WHEAT Trial during a time period when the SWAT is active at their site

Exclusion Criteria:

Infant or family ineligible for participation in the WHEAT International Trial

Parent(s)/primary caregiver(s) not approached for WHEAT Trial participation (e.g., missed recruitment window, language barriers not addressed by materials, medical instability of infant or family)

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 787 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Opt-in Rate for the WHEAT International Trial | Baseline (When the family is approached for the Study Participation - Within first two weeks of life))
  The proportion of families approached for participation in the WHEAT International Trial who provide consent (or do not opt out, depending on the site's consent model) for their infant to be enrolled.

SECONDARY OUTCOMES:
Trial Withdrawal Rate (Post-Randomization) | Birth to 40 weeks Post Menstrual Age (From enrollment until study completion)
  The proportion of enrolled participants who withdraw from the WHEAT International Trial after randomization.
Parental Comprehension of Trial-Specific Details | Baseline (Once family makes the consent decision - Within first two weeks of life)
  Degree to which parents understand key elements of the WHEAT International Trial, assessed via a brief questionnaire co-designed with a parent-partner group.
Parental Experience with the Consent Process | Baseline (Once family makes the consent decision - Within first two weeks of life)
  Parents' perceptions of the clarity, helpfulness, and adequacy of the information provided during the consent process, collected via a brief, co-designed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Balpreet Singh, Principal Investigator — IWK Health
Locations (15):
- Canada (15):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - BC Women's Hospital and Health Centre, Vancouver, British Columbia
  - Dr. Everett Chalmers, Fredericton, New Brunswick
  - Moncton Hospital, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Janeway Children's Health and Rehabilitation Centre, Saint Johns, NFLD
  - IWK Health, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital/CHEO, Ottawa, Ontario
  - Mount Sinai, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Centre hospitalier de l'Université Laval, Laval, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lawrence LM, Bishop A, Curran J. Integrated Knowledge Translation with Public Health Policy Makers: A Scoping Review. Healthc Policy. 2019 Feb;14(3):55-77. doi: 10.12927/hcpol.2019.25792. PMID 31017866
- [Background] Korstjens I, Moser A. Series: Practical guidance to qualitative research. Part 4: Trustworthiness and publishing. Eur J Gen Pract. 2018 Dec;24(1):120-124. doi: 10.1080/13814788.2017.1375092. Epub 2017 Dec 5. PMID 29202616
- [Background] Elo S, Kyngas H. The qualitative content analysis process. J Adv Nurs. 2008 Apr;62(1):107-15. doi: 10.1111/j.1365-2648.2007.04569.x. PMID 18352969
- [Background] Ouyang Y, Karim ME, Gustafson P, Field TS, Wong H. Explaining the variation in the attained power of a stepped-wedge trial with unequal cluster sizes. BMC Med Res Methodol. 2020 Jun 24;20(1):166. doi: 10.1186/s12874-020-01036-5. PMID 32580698
- [Background] Voldal EC, Hakhu NR, Xia F, Heagerty PJ, Hughes JP. swCRTdesign: An RPackage for Stepped Wedge Trial Design and Analysis. Comput Methods Programs Biomed. 2020 Nov;196:105514. doi: 10.1016/j.cmpb.2020.105514. Epub 2020 May 21. PMID 32554025
- [Background] Synnot A, Ryan R, Prictor M, Fetherstonhaugh D, Parker B. Audio-visual presentation of information for informed consent for participation in clinical trials. Cochrane Database Syst Rev. 2014 May 9;2014(5):CD003717. doi: 10.1002/14651858.CD003717.pub3. PMID 24809816
- [Background] Ballard HO, Shook LA, Desai NS, Anand KJ. Neonatal research and the validity of informed consent obtained in the perinatal period. J Perinatol. 2004 Jul;24(7):409-15. doi: 10.1038/sj.jp.7211142. PMID 15152271
- [Background] Wilman E, Megone C, Oliver S, Duley L, Gyte G, Wright JM. The ethical issues regarding consent to clinical trials with pre-term or sick neonates: a systematic review (framework synthesis) of the empirical research. Trials. 2015 Nov 4;16:502. doi: 10.1186/s13063-015-0957-x. PMID 26537492
- [Background] Dahav P, Sjostrom-Strand A. Parents' experiences of their child being admitted to a paediatric intensive care unit: a qualitative study-like being in another world. Scand J Caring Sci. 2018 Mar;32(1):363-370. doi: 10.1111/scs.12470. Epub 2017 Aug 22. PMID 28833379
- [Background] Obeidat HM, Bond EA, Callister LC. The parental experience of having an infant in the newborn intensive care unit. J Perinat Educ. 2009 Summer;18(3):23-9. doi: 10.1624/105812409X461199. PMID 20514124
- [Background] Al Maghaireh DF, Abdullah KL, Chan CM, Piaw CY, Al Kawafha MM. Systematic review of qualitative studies exploring parental experiences in the Neonatal Intensive Care Unit. J Clin Nurs. 2016 Oct;25(19-20):2745-56. doi: 10.1111/jocn.13259. Epub 2016 Jun 3. PMID 27256250